CLINICAL TRIAL: NCT00061438
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Study on the Use of Prophylactic Meropenem Therapy in Subjects With Severe Acute Necrotizing Pancreatitis
Brief Title: A Study to Determine if Antibiotics Prevent Infection in the Pancreas of Patients Where Part of the Pancreas Has Died
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3591IL/0089; 89
Record Dates: First submitted 2003-05-27; First posted 2003-05-28 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Pancreatitis, Acute Necrotizing
Keywords: non-infected necrotizing pancreatitis; pancreatic infection; peripancreatic infection
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing | interventions — Meropenem

INTERVENTIONS:
Drug: meropenem

SUMMARY:
This is a research study in patients having a condition known as necrotizing pancreatitis. This is inflammation of the pancreas (an intestinal organ which assists with digestion) that has resulted in the damage and death of some pancreatic tissue. This damaged pancreatic tissue may develop a bacterial infection, which can cause further -sometimes very serious- health problems.

It may be possible to prevent or delay infection by giving 'prophylactic' antibiotics (that is - to provide protection before any infection starts). However, it is not certain that this antibiotic therapy will be successful.

This study is being carried out to see whether the antibiotic 'Meropenem' (which is also known as MERREM I.V.) provides protection from developing a pancreatic infection. This will be done by comparing the progress of patients who receive meropenem with those who receive a non-active placebo solution (a solution that does not contain any active medication).

Meropenem or placebo would be given in addition to the standard treatment received for pancreatitis.

It is not known if meropenem will help prevent infections associated with necrotizing pancreatitis.

Approximately 240 patients will take part in this study.

Study participation will be carried out for up to 6 weeks, and patients will receive the study treatment up to a maximum of 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of necrotizing pancreatitis within 120 hours following onset of symptoms/first reported symptoms.
* Primary diagnosis to be confirmed by contrast-enhanced CT evidence of 30% necrosis of the pancreas.
* Or if > or equal to 30% necrosis is not present or cannot be confirmed, a contrast enhanced CT scan showing extensive or multiple pancreatic fluid collections and pancreatic edema (Balthazar Grade E) with either C-reactive protein (CRP). 120 mg/L or a MOD score of > 2 is acceptable.

Exclusion Criteria:

* Received an investigational drug or device within 30 days prior to entering study.
* Received > 48 hours of antibiotic therapy between onset of symptoms of pancreatitis and diagnosis of necrotizing pancreatitis.
* The subject has known or suspected anaphylactic or other type 1 (immediate) hypersensitivity reactions to cephalosporins, penicillins or carbapenems.
* The subject is receiving, or will require, probenecid therapy.
* The subject is neutropenic (absolute neutrophil count < 1000/mm 3).
* The subject has cirrhosis, severity of Child's grade C.
* There is not a commitment on the part of the clinical care team, the subject, or the subject's family to full, aggressive support including operative intervention if needed.
* The subject is a pregnant and/or nursing female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2003-02; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AntiInfection Medical Science Director, MD, Study Director — AstraZeneca
Locations (11):
- United States (9):
  - Research Site, San Francisco, California
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Newark, New Jersey
  - Research Site, New York, New York
  - Research Site, Seattle, Washington
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec